CLINICAL TRIAL: NCT03668197
Title: Children Peritonitis Ecology at CHU de Rennes - (IIAPEDIA)
Acronym: IIAPEDIA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3086_IIAPEDIA
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: microbiological analysis — microbiological analysis of the peritoneal fluid

SUMMARY:
The main objectif is assess the germs (species + antibiograms) implicated in children intra-abdominal infections (community acquired or nosocomial ) at CHU de Rennes.

ELIGIBILITY:
Inclusion Criteria:

* Children between 0 and 18 years old
* Intra-abdominal infection with and indication for surgery or radiologically guided drainage.
* No opposition from the child or his parents

Exclusion Criteria:

* No microbiological sampling.
* Primitive peritonitis (Spontaneous bacterial peritonitis, peritonitis during peritoneal dialysis)

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Intra-abdominal infection and indication for surgery or radiologically guided drainage
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-01-26 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Blood Culture | 2 weeks after inclusion
  Ecology (germs resistance profile)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France